CLINICAL TRIAL: NCT01533051
Title: Phase IV Study of Durability of Anti-viral Therapy in Patients With Chronic Hepatitis B
Brief Title: Prospective Observational Cohort Study for the Durability of Anti-viral Therapy in Patients With Chronic Hepatitis B
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, Sang Hoon Ahn, Associate Professor, Yonsei University
Other Study IDs: Quit Anti-viral therapy
Record Dates: First submitted 2012-02-07; First posted 2012-02-15 (Estimated); Last update posted 2012-05-08 (Estimated); Status verified 2012-05

CONDITIONS: Chronic Hepatitis B
Keywords: Chronic hepatitis B; Nucleos(t)ide analogue; Antiviral treatment; Korea
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Initially, 30ml of heparinized peripheral blood will be obtained from each subjects. After then, 10ml of heparinized peripheral blood will be additionaly obtained at every 3 months follow-up visit.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Chronic hepatitis B

SUMMARY:
The aim of this study is to investigate the off-treatment sustained virological and biochemical response in chronic hepatitis B patients following the guideline by the Asian Pacific Association for the Study of the Liver (APASL) in Korea.

DETAILED DESCRIPTION:
In the recommendation by the Asian PAcific Association for the Study of the Liver(APASL), antiviral drug is recommended to stop when HBeAg seroconversion has developed for more than 6 months among HBeAg-positive patietns. For HBeAg-negative patients, the APASL consensus recommended stopping anti-viral treatment when HBV DNA remained undetectable for three separates occasion 6 months apart. Nontheless, approximately 25% to 50% of the patients still develop hepatitis relapse after stopping anti-viral therapy even if these recommendations are followed. In this study, the investigators aimed to investigated the off-treatment sustained response in chronic hepatitis B parients following the stopping anti-viral treatment guideline in Korea.

ELIGIBILITY:
Inclusion Criteria:

* More than 20 years old
* Chronic hepatitis B patients under anti-viral therapy

  1. In HBeAg-positive patient; if HBeAg seroconversion with undetectable HBV DNA is documented on two separate occasions at least 6 months
  2. In HBeAg-negative patient; if undetectable HBV DNA has been documented on three separate occasions 6 months apart

Exclusion Criteria:

* Patients who had chronic liver disease due to hemochromatosis, autoimmune hepatitis, drug-induced hepatitis, or thalassemia
* Patients who suffered from other chronic medical condition

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic Hepatitis B patients under anti-viral therapy
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2012-02; Primary Completion 2015-03 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Sustained virological response after stopping anti-viral treatment | Up to 3 years
  The proportion of patients with sustained virological response after stopping anti-viral treatment

CONTACTS AND LOCATIONS:
Overall Officials: Sang Hoon Ahn, MD, PhD, Study Chair — Department of Internal Medicine, Yonsei Universtiy College of Medicine
Locations (1):
- Sang Hoon Ahn, Seoul, South Korea